CLINICAL TRIAL: NCT05441956
Title: A Dose Escalation and Expansion Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TGRX-326 Monotherapy for the Treatment of Advanced ALK-positive or ROS1-positive Non-Small Cell Lung Cancer
Brief Title: TGRX-326 Chinese Phase I for Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-326-1001
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TGRX-326 (Experimental): Subjects to be treated with the investigational drug TGRX-326
  Interventions: Drug: TGRX-326

INTERVENTIONS:
Drug: TGRX-326 — Participants are given TGRX-326 tablets orally at one of the dose levels as pre-determined.

SUMMARY:
This trial is a multi-center, single-arm, open-label, Phase I clinical trial in 3 phases: dose escalation phase, dose expansion phase and indication expansion phase, which will explore the safety, tolerability, PK and preliminary efficacy of TGRX-326 in patients with ALK-positive or ROS1-positive advanced NSCLC.

DETAILED DESCRIPTION:
This is the first-in-human trial with TGRX-326 which aims to evaluate the safety profile and preliminary efficacy profile in patients with ALK-positive or ROS1-positive advanced NSCLC. The primary purpose of this study is to evaluate the safety profile of TGRX-326, including determination of the maximal tolerated dose (MTD) and recommended phase II dose (RP2D), and other safety measures of the investigational drug, such as adverse events and abnormal clinical outcomes. Preliminary efficacy profiles of TGRX-326 is also evaluated according to RECIST Version 1.1. The safety, tolerability and efficacy profiles, along with pharmacokinetic analysis, will be assessed together to determine the optimal dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

* Willing to follow the treatment protocol and visit schedule, and participate in the study with the ICF signed;
* ≥ 18 years of age on the day of ICF signing, regardless of gender.
* Diagnosis of ALK-positive or ROS1-positive advanced NSCLC by histopathology or cytology in a Grade-A tertiary hospital or central laboratory.
* Provision of the following information: archived tissue samples and/or fresh tumor tissue samples obtained during the screening period for biomarker detection; previous biomarker detection results from a Grade-A tertiary hospital (exempt from the above-mentioned biomarker detection); previous NGS results; the consent of medical monitors for the participation of subjects who fail to provide tumor tissue samples (e.g., samples are exhausted due to previous diagnostic tests but high clinical risk may be brought about by re-puncture, etc.).
* Metastases to central nervous system (CNS) with the following conditions met: a. asymptomatic: no current need for corticosteroid therapy, or only stable dose or a dose reduced to ≤ 10 mg of prednisone (QD) or equivalent required; or b. past diagnosis, treatment completed, complete recovery from acute effects of radiation therapy or surgery prior to the first dose, discontinuation of corticosteroid therapy for these metastases for at least 4 weeks, and neurologically stable;
* Drug discontinuation for ≥ 5 half-lives prior to the first dose for subjects previously treated with a targeted therapy (e.g., ALK or ROS1 inhibitors);
* At least one measurable (longest diameter for non-lymph nodes: ≥ 10 mm; shortest diameter for lymph nodes: ≥ 15 mm) target lesion (a previously irradiated lesion cannot be regarded as a target lesion unless it is significantly progressive) according to criteria in RECIST version 1.1;
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0-1 point in dose escalation and dose expansion phases; 0-2 points in indication expansion phase;
* Recovery from any AEs associated with prior surgery and cancer therapy (to ≤ Grade 1), with the following exceptions: a. alopecia; b. pigmentation; c. long-term toxicity due to radiotherapy that, in the judgment of the investigator, is not recoverable; d. Grade 2 and below neurotoxicity due to platinum; e. hemoglobin within the range of 90-100 g/L (inclusive);
* Adequate bone marrow, liver, kidney, coagulation and pancreatic functions;
* Expected survival ≥ 3 months;
* Willing to take effective contraceptive measures (for men of reproductive potential and women of reproductive age only) from ICF signing to 6 months after administration of the investigational drug. Women of reproductive age include women in perimenopause and within 2 years after menopause. Those women must have a negative pregnancy test ≤ 7 days prior to the first dose of the investigational drug.

Exclusion Criteria:

* Previous use of any third-generation ALK inhibitors or second-generation ROS1 inhibitors other than TGRX-326.
* Known hypersensitivity to any of the active ingredients or excipients of TGRX-326; an identified history of allergy to protein-based drugs; a history of atopic allergy (asthma, rheumatism, eczematous dermatitis); previous history of other severe allergic reactions that makes himself/herself unsuitable for TGRX-326 treatment in the judgment of the investigator;
* Having another type of cancer except for lung cancer, excluding malignant tumors including cervical cancer in situ and non-melanoma skin cancer that have been curatively treated and have not recurred within 5 years;
* Having previously received antibodies or pharmacotherapy against T cell costimulation or immune checkpoint pathways, including but not limited to anti-programmed cell death protein 1 (anti-PD-1), anti-programmed cell death protein ligand 1 (anti-PD-1), anti-programmed cell death protein ligand 2 (anti-PD-L2), anti-cluster of differentiation 137 (anti-CD137) antibody or anti-cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody;
* Major surgery within 4 weeks prior to the first dose. Minor surgery such as infusion port placement is not listed in the exclusion criteria, but sufficient time is required to achieve adequate wound healing;
* Spinal cord compression, unless the subject achieves significant pain control with treatment and full recovery of neurological function within 4 weeks prior to the first dose.
* Abnormal gastrointestinal function, including the inability to take oral drugs, the need for intravenous nutrition, previous surgical operations (including total gastrectomy or gastric band surgery) that affect absorption, active inflammatory gastrointestinal diseases, chronic diarrhea, symptomatic Diverticular disease, treatment of active peptic ulcer disease or malabsorption syndrome within the past 6 months;
* History of active pneumonia or interstitial pneumonia, or radiation or drug-induced lung disorder on CT at screening. Radiation pneumonia patients without clinical symptoms 3 months after radiotherapy are allowed to be enrolled;
* Cardiac insufficiency, including but not limited to left ventricular ejection fraction (LVEF) < 50%, history of congestive cardiac failure, ventricular arrhythmia requiring treatment, hypokalemia, hereditary long QT syndrome, or history of myocardial infarction or unstable angina pectoris within 6 months before screening; ≥ Class 2 heart failure in New York Heart Association Classification;
* Abnormal and clinically significant QTc on ECG (> 450 msec [male] or QTc > 470 msec [female] at rest); concomitant use of any drug known to prolong QT interval and cause torsades de pointes;
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) after drug treatment;
* Susceptibility to acute pancreatitis (e.g., uncontrolled hyperglycemia, current gallstones) as judged by the investigator one month prior to the first dose;
* Severe or uncontrolled systemic diseases (such as unstable or uncompensated respiratory, cardiac, hepatic or renal diseases) causing expected intolerance to the investigational drug as judged by the investigator;
* Use within 14 days before first dose or expected concomitant use during the treatment period of drugs that pose risk of QTC interval prolongation and/or ventricular tachycardia;
* Use of any systemic antineoplastic therapies within 28 days prior to the first dose of trial drug (included if TGRX-326 is allowed within 28 days after the systemic antineoplastic therapy, as assessed by the investigator), including systemic chemotherapy, immunotherapy (physiological replacement dose of glucocorticoids [prednisone or equivalent < 10 mg/day] is allowed, excluding antibodies or drugs against T-cell costimulation or immune checkpoint pathways).
* Treatment with radiotherapy or Chinese herbal medicine or Chinese patent medicine for antineoplastic therapies within 14 days prior to the first dose.
* Subjects who have withdrawn from a low dose group due to disease progression and then have been re-enrolled in a higher dose group do not have limited washout period for systemic antineoplastic therapies prior to re-administration of the investigational drug;
* Clinically significant active bacterial, fungal or viral infections, including a positive result for hepatitis B surface antigen and HBV; one or more positive results for hepatitis C antibody, treponema pallidum antibody, or HIV antibody; the presence of any uncontrolled infection.
* Use of strong CYP3A4 inducers or inhibitors or CYP3A4 substrates with a narrow therapeutic window within two weeks prior to the first dose of the investigational drug;
* Pregnant and breastfeeding female;
* Women of childbearing age who are unwilling or unable to use acceptable methods for contraception during the entire treatment period in the trial and within 6 months after the last dose of the investigational drug (women of childbearing age include: any one with menarche, and those who have not received successful artificial sterilization [hysterectomy, bilateral fallopian tube ligation, or bilateral oophorectomy] or premenopausal women); a fertile male patient who is unwilling or unable to take effective contraceptive measures, and whose partner is a woman of childbearing age;
* Being involved in other clinical studies; less than 4 weeks from the end of the previous clinical study to the first dose of the investigational drug or 5 half-lives of the previous drug, whichever is shorter;
* Any mental or cognitive disorders which may limit subjects' understanding and implementation of the informed consent form;
* Other situations, such as poor compliance, which are considered by the investigator not to be suitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) | At end of Cycle 1 (each cycle is 21 days) when the probability of DLT of a dose level is higher than 33%
  To determine the MTD of TGRX-326 in NSCLC patients
Recommended phase II dose (RP2D) | At completion of the dose expansion study, an average of 1 year
  To determine the RP2D of TGRX-326 in NSCLC patients for Phase II
Safety profile (DLT) | Collect during Cycle 1 (each cycle is 21 days)
  To record and analyse subjects with dose-limiting toxicities (DLTs)
Safety profile (AEs/SAEs) | Through completion of the study, an average of 1.5 years
  To record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Plasma Cmax | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Cmax of TGRX-326 as measured in plasma
Plasma Tmax | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Tmax of TGRX-326 as measured in plasma
T1/2 | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Half life of TGRX-326 as measured in plasma
Plasma AUCinf | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  AUCinf of TGRX-326 as measured in plasma
Plasma Cmin | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Cmin of TGRX-326 as measured in plasma
Plasma AUCss | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  AUCss of TGRX-326 as measured in plasma
Plasma Cmax,ss | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Cmax at steady state of TGRX-326 as measured in plasma
Plasma Tmax,ss | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Tmax at steady state of TGRX-326 as measured in plasma
CL | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Clearance of TGRX-326 as measured in plasma
Vd | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Volume of distribution of TGRX-326 as measured in plasma
Plasma T1/2,ss | Day1/3 of single-dose period; Day1/8/15 of Cycle 1; Day1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  T1/2 at steady state of TGRX-326 as measured in plasma
ORR | At screening, Day 1 of every other cycle starting from Cycle 3, and Day 1 of every 4 cycles starting Cycle 17 (each cycle is 21 days)
  Objective response rate (ORR) as the percentage of patients achieving a CR or PR
IC-ORR | At screening, Day 1 of every other cycle starting from Cycle 3, and Day 1 of every 4 cycles starting Cycle 17 (each cycle is 21 days)
  Intracranial objective response rate (IC-ORR) as the percentage of patients achieving an intracranial CR or PR among those with confirmed intracranial lesions
DCR | At screening, Day 1 of every other cycle starting from Cycle 3, and Day 1 of every 4 cycles starting Cycle 17 (each cycle is 21 days)
  Disease control rate (DCR) as the percentage of patients who achieve a response (PR + CR) and stable disease (SD) after the treatment
IC-DCR | At screening, Day 1 of every other cycle starting from Cycle 3, and Day 1 of every 4 cycles starting Cycle 17 (each cycle is 21 days)
  Intracranial disease control rate (IC-DCR) as the percentage of patients achieving an intracranial response (PR + CR) and a stable disease (SD) after the treatment among those with confirmed intracranial lesions
DOR | At screening, Day 1 of every other cycle starting from Cycle 3, and Day 1 of every 4 cycles starting Cycle 17 (each cycle is 21 days)
  Duration of response (DOR) as the length of time from the first confirmation of CR or PR until the date of the first occurrence of PD or death, applicable to subjects achieving a response only
IC-DOR | At screening, Day 1 of every other cycle starting from Cycle 3, and Day 1 of every 4 cycles starting Cycle 17 (each cycle is 21 days)
  Intracranial duration of response (IC-DOR) as the length of time from the first confirmation of intracranial CR or intracranial PR until the date of the first occurrence of PD or death, applicable to subjects achieving an intracranial response only

OTHER OUTCOMES:
Cmax, CSF | Day 1/3 of single-dose period; Day 1/8/15 of Cycle 1; Day 1 of Cycle 2-5, Day 1 of every other cycle starting from Cycle 7; Day 1 of every 4 cycles starting from Cycle 17 (each cycle is 21 days)
  Cmax of TGRX-326 as measured in cerebral-spinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao S, Zhou H, Yang N, Wang Z, Jin W, Ma Y, Xue J, Li X, Liu Y, Meng R, Zhou J, Cheng Y, Wang Y, Yu Z, Cao Y, Zhao Y, Huang Y, Fang W, Zhang Y, Hong S, Wu B, Shi Y, Cao J, Xu M, Zhang X, Hu L, Peng B, Yang Y, Zhang L, Zhao H. Safety, Efficacy, and Biomarker Analysis of Deulorlatinib (TGRX-326) in Anaplastic Lymphoma Kinase-Positive NSCLC: A Multicenter, Open-Label, Phase 1/1b Trial. J Thorac Oncol. 2025 Jun;20(6):750-762. doi: 10.1016/j.jtho.2024.11.010. Epub 2024 Nov 15. PMID 39551469